CLINICAL TRIAL: NCT00725478
Title: Stabilization on, or Change-over to the Non-ergot Dopamine Agonist Piribedil in Patients With Morbus Parkinson - a Post Marketing Surveillance Study in Parkinson Clinic Ambulances and Larger Private Practices.
Brief Title: SEDPARK1: Safety and Efficacy Study With the Non-ergot Dopamine-agonist Piribedil in Parkinson's Disease
Acronym: PIR-001/K
Status: Completed | Type: Observational
Sponsor: Desitin Arzneimittel GmbH (Industry)
Responsible Party: Dr. Martina Wangemann, Desitin Arzneimittel GmbH
Other Study IDs: PIR-001/K
Record Dates: First submitted 2008-07-28; First posted 2008-07-30 (Estimated); Last update posted 2010-03-31 (Estimated); Status verified 2008-07

CONDITIONS: Parkinson's Disease
Keywords: Piribedil (trade name: CLARIUM); non-ergot dopamine agonist; Morbus Parkinson; Tolerability; Efficacy; Post Marketing Surveillance
MeSH Terms: conditions — Parkinson Disease | interventions — Piribedil

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Piribedil

SUMMARY:
The aim of the non-interventional Post Marketing Study is to investigate the use of the non-ergot dopamine agonist piribedil (trade name: CLARIUM) in mono- and combination therapy in patients with Morbus Parkinson. Tolerability and course of the disease or change of parkinsonian symptoms during stabilisation on, or change over from other dopamine agonists will be documented under routine conditions. Piribedil should be prescribed according to its marketing authorisation by the responsible neurologist.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients 18 years and older.
* Indication: Morbus Parkinson.
* Treatment with piribedil for the first time.
* Monotherapy with piribedil.
* Combination therapy with L-Dopa (from the beginning or secondary) and/or in combination with other antiparkinsonian drugs.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Morbus Parkinson who require therapy with dopamine agonists.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
to monitor use in real practice including adverse events on piribedil | 3 months

SECONDARY OUTCOMES:
Efficacy | 3 months

REFERENCES:
- [Background] Castro-Caldas A, Delwaide P, Jost W, Merello M, Williams A, Lamberti P, Aguilar M, Del Signore S, Cesaro P; Parkinson-Control Study Group. The Parkinson-Control study: a 1-year randomized, double-blind trial comparing piribedil (150 mg/day) with bromocriptine (25 mg/day) in early combination with levodopa in Parkinson's disease. Mov Disord. 2006 Apr;21(4):500-9. doi: 10.1002/mds.20750. PMID 16267842
- [Background] Rascol O, Dubois B, Caldas AC, Senn S, Del Signore S, Lees A; Parkinson REGAIN Study Group. Early piribedil monotherapy of Parkinson's disease: A planned seven-month report of the REGAIN study. Mov Disord. 2006 Dec;21(12):2110-5. doi: 10.1002/mds.21122. PMID 17013922
- [Background] Rascol O, Pathak A, Bagheri H, Montastruc JL. Dopaminagonists and fibrotic valvular heart disease: further considerations. Mov Disord. 2004 Dec;19(12):1524-5. doi: 10.1002/mds.20328. No abstract available. PMID 15515031